CLINICAL TRIAL: NCT06022289
Title: Safety and Efficacy of Pemigatinib in the Treatment of Advanced Pan Solid Tumors With FGF/FGFR Alterations: An Open, Single-arm, Prospective Phase II Trial
Brief Title: Pemigatinib for FGF/FGFR Alterations Advanced Pan Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pemigatinib for Pan-cancer
Record Dates: First submitted 2023-08-19; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumor; FGF Receptor Gene Mutation; FGF Amplification; FGF Receptor Gene Family Rearrangement; FGF Receptor Gene Translocation
Keywords: Solid Tumor; FGFR; Pemigatinib
MeSH Terms: interventions — pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monotherapy or combination therapy based on Pemigatinib (Experimental): Pemigatinib will be treated according to the treatment plan of 2 weeks of administration/1 week of discontinuation, with oral administration of 1 capsule, 13.5mg, QD, and a cycle of 21 days. Meanwhile, the molecular testing results of the patient are analyzed and interpreted by the MTB team, and appropriate combination therapy(Pemigatinib+) strategies are proposed based on the patient's previous treatment history, physical condition, drug accessibility, and economic status.
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — Pemigatinib will be treated according to the treatment plan of 2 weeks of administration/1 week of discontinuation, with oral administration of 1 capsule, 13.5mg, QD, and a cycle of 21 days. Meanwhile, the molecular testing results of the patient are analyzed and interpreted by the MTB team, and appropriate combination therapy(Pemigatinib+) strategies are proposed based on the patient's previous treatment history, physical condition, drug accessibility, and economic status.
  Other Names: INCB05482

SUMMARY:
The purpose of this clinical trial is to demonstrate safety and efficacy of Pemigatinib in the treatment of advanced pan solid tumor patients with FGF/FGFR alterations.

DETAILED DESCRIPTION:
This study is a prospective, single arm, phase II clinical study. Patients with advanced solid tumors who had previously failed standard treatment and had FGFR1-3 alterations were selected and included in this study after signing the informed consent form and meeting the inclusion criteria. The patient will receive oral treatment with pemitinib (13.5 mg QD, administered for 2 weeks/discontinued for 1 week). Before assessment for eligibility, patients were prescreened centrally for FGF/FGFR status using massively parallel DNA sequencing.Patients who already had an FGF/FGFR status report based on local assessment (Clinical Laboratory Improvement Amendments [CLIA]-certifed) or an existing MTB approved report were also included. The subjects will continue treatment until disease progression or intolerable toxicity occurs. During the treatment process, clinical tumor imaging evaluation was conducted according to RECIST v1.1, every 6 weeks (± 7 days), and every 9 weeks (± 7 days) after 48 weeks. Use NCI-CTCAE 5.0 for safety assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old; Gender unlimited
2. Late stage, recurrent, or metastatic solid tumors confirmed by histology or cytology as unresectable by surgery.
3. According to RECIST v1.1, there is at least one measurable lesion.
4. Histological confirmation of FGFR1-3 alterations, including but not limited to amplification, mutation, fusion/rearrangement, etc.
5. After standard treatment, the disease progresses, becomes intolerable, or standard treatment is ineffective, or there is no standard treatment plan.
6. Has not previously used small molecule multi target inhibitors targeting the FGFR pathway (including arotinib, lenvatinib, sorafenib, apatinib, etc.).
7. ECOG physical fitness status is 0-1.
8. Expected survival time>3 months.
9. Sufficient organ function is required for the subject to meet the following laboratory indicators:

   1. In the past 14 days without using granulocyte colony stimulating factor, the absolute value of neutrophils (ANC) ≥ 1.5x10^9/L.
   2. Platelets ≥ 100 without blood transfusion in the past 14 days × 10^9/L.
   3. In the absence of blood transfusion or use of erythropoietin within the past 14 days, hemoglobin>9g/dL.
   4. Total bilirubin ≤ 1.5 × Upper limit of normal value (ULN). Or total bilirubin>ULN but direct bilirubin ≤ ULN.

      5) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) are ≤ 2.5 × ULN (ALT or AST ≤ 5 allowed for patients with liver metastasis) × ULN).

      6) Blood creatinine ≤ 1.5 × ULN and creatinine clearance rate (calculated using Cockcroft Fault formula) ≥ 50 ml/min.

      7) Good coagulation function, defined as international standardized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN. If the subject is undergoing anticoagulant therapy, as long as the PT is within the prescribed range of anticoagulant drugs, it is sufficient.
10. For female subjects of childbearing age, they should undergo a urine or serum pregnancy test with a negative result within 3 days before receiving the first study drug administration (day 1 of cycle 1). If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required. Non reproductive age women are defined as those who have undergone at least one year of menopause or have undergone surgical sterilization or hysterectomy.
11. If there is a risk of conception, all subjects (whether male or female) are required to use contraceptive measures with an annual failure rate of less than 1% throughout the entire treatment period until 120 days after the last study drug administration (or 180 days after the last chemotherapy drug administration).

Exclusion criteria:

1. Diagnosed within 5 years prior to the first administration as other malignant diseases outside of the current enrollment diagnosis (excluding basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or carcinoma in situ after radical resection).
2. Previously received selective FGFR inhibitor treatment.
3. Those who have received any other study drug treatment or participated in intervention clinical studies within 28 days before the first administration. Or received anti-tumor drug treatment (including Chinese herbal medicine with anti-tumor indications) within 28 days before the first use of the study drug.
4. Not fully recovered from toxicity and/or complications caused by any intervention measures before starting treatment (i.e. ≤ level 1 or reaching baseline, excluding fatigue or hair loss).
5. Symptomatic central nervous system metastasis and/or cancerous meningitis are known to exist. For brain metastasis subjects who have previously received treatment, if their condition is stable (there is no evidence of imaging progression within at least 4 weeks before the first administration of the trial treatment), repeated imaging examinations confirm no evidence of new brain metastasis or enlargement of existing brain metastasis lesions, and steroid treatment is not required at least 14 days before the first administration of the trial treatment, they can participate in the trial. This exception does not include cancerous meningitis, which should be excluded regardless of its clinical stability.
6. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
7. The following laboratory parameters are abnormal:

   1. Serum phosphate>ULN.
   2. Serum calcium exceeds the normal range, or when serum albumin exceeds the normal range, the corrected calcium concentration of serum albumin exceeds the normal range.
   3. Potassium level<lower limit of normal value. Potassium levels can be corrected through supplementation during screening.
8. Known history of human immunodeficiency virus (HIV) infection or confirmed positive immune test results.
9. Severe infections with active or poorly controlled clinical conditions.
10. Chest fluid, ascites, or pericardial effusion with obvious clinical symptoms that require drainage treatment.
11. Individuals infected with acute or chronic active hepatitis B or hepatitis C, with hepatitis B virus (HBV) DNA>2000IU/ml or 10^4 copies/ml. Hepatitis C virus (HCV) RNA>10^3 copies/ml. Hepatitis B surface antigen (HbsAg) and anti HCV antibody were positive at the same time. Those who have undergone nucleotides based antiviral treatment and fall below the above standards can be enrolled in the group.
12. Clinically significant or uncontrolled heart diseases, including unstable angina pectoris, acute myocardial infarction occurring within 6 months prior to first administration, New York Heart Association Class III/IV congestive heart failure, and uncontrolled arrhythmia (allowing subjects with pacemakers or atrial fibrillation and good heart rate control).
13. There are ECG changes or medical histories that researchers believe have clinical significance. Screening QTcF interval>480 ms, for subjects with indoor conduction block (QRS interval>120 ms), JTc interval can be used instead of QTc interval (if JTc is used instead of QTc, JTc must be ≤ 340 ms).
14. Uncontrolled hypertension, with systolic blood pressure>160 mmHg or diastolic blood pressure>100 mmHg after optimal medical treatment, hypertension crisis or history of hypertensive encephalopathy.
15. Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh B grade or more severe cirrhosis.
16. Has undergone major surgical procedures (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of study treatment or is expected to require major surgery during the study treatment period.
17. Toxicity and/or major surgical complications have not yet fully recovered before starting treatment.
18. Pregnant or lactating women, or subjects who are expected to conceive or give birth during the study period from screening visits to completion of safety follow-up visits (male subjects up to 90 days after last administration).
19. Received radiotherapy within 4 weeks prior to the first administration of the study drug. The radiation related toxicity of the subject must have fully recovered, and corticosteroid treatment is not required. It is confirmed that radiation pneumonia has been ruled out. For palliative radiotherapy for non-CNS diseases, a 2-week washout period is allowed.
20. Have a history of systemic electrolyte metabolism imbalance caused by calcium and phosphorus metabolism disorders or accompanied by soft tissue ectopic calcification (excluding skin, kidney, tendon, or vascular calcification caused by injuries, diseases, and advanced age without systemic electrolyte metabolism imbalance).
21. Corneal or retinal diseases confirmed to have clinical significance through ophthalmic examination.
22. Any potent CYP3A4 inhibitor (see Appendix A for details) or inducer has been used within 14 days or 5 half-lives before the first administration of the study drug, whichever is shorter. Allow external use of ketoconazole.
23. It is known that there is an allergic reaction to Pemigatinib or its research drug excipients.
24. Unable or unwilling to swallow Pemigatinib or suffering from significant digestive system diseases that may interfere with absorption, metabolism, or excretion.
25. The subject has a history of vitamin D deficiency and needs to supplement vitamin D beyond physiological levels (excluding vitamin D dietary supplements).
26. Other acute or chronic diseases, mental illnesses, or abnormal laboratory test values that may lead to increased risk of study participation or drug administration, or interference with the interpretation of study results, and the inclusion of patients as ineligible to participate in this study based on the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival 2/Progression-free Survival 1(PFS2/PFS1) | Through study completion, an expected average of 1 year.
  The progression free survival (PFS1) after the most recent treatment before enrollment is defined as the progression of the disease from the most recent treatment before enrollment.The progression free survival period (PFS2) after enrollment is defined as the time from matched targeted therapy or unmatched therapy to disease progression or death.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Through study completion, an expected average of 1 year.
  The proportion of patients whose tumor volume is reduced to 30% and can be maintained for more than 4 weeks,Based on RECIST criteria v1.1.
Progression-free Survival (PFS) | The last subject completes at least 24 weeks of follow-up (or disease progression).
  The time from the beginning of the patient's treatment to the disease progression or death for any reason.Based on RECIST criteria v1.1.
Disease control rate (DCR) | Through study completion, an expected average of 1 year.
  The DCR was defined as SD, PR or CR according to RECIST criteria v1.1.
Overall survival(OS) | Through study completion, an expected average of 2 years.
  The time from the patient receiving treatment to the death of the patient for any reason,OS evaluated according to RECIST v1.1.
Duration of Response(DOR) | Through study completion, an expected average of 1 year.
  Duration of Response,from the first time the evaluation results meet CR or PR criteria to the observation of PD or death.
Adverse events(AEs） | Through study completion, an expected average of 2 years.
  Include Treatment emerge adverse events, treatment related adverse events and serious adverse events,AEs evaluated according to NCI-CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: HaiTao Wang, Ph.D, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical University Second Hospital, Tianjin, Tianjin Municipality, China